CLINICAL TRIAL: NCT04947722
Title: The PREVENT Trial: a Pragmatic Cluster Randomized Controlled Trial of a Multifaceted Fracture Prevention Model for Long-term Care
Acronym: PREVENT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Alexandra Papaioannou, Executive Director, GERAS Centre for Aging Research, Hamilton Health Sciences, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 13622
Record Dates: First submitted 2021-06-24; First posted 2021-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Fracture; Fractures, Hip; Osteoporosis
Keywords: Long-Term Care; Fracture Risk; Falls; Knowledge Translation
MeSH Terms: conditions — Fractures, Bone; Hip Fractures; Osteoporosis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PREVENT Program (Experimental): PREVENT model
  Interventions: Behavioral: PREVENT Program
- Control Group (No Intervention): Residents in homes allocated to the control group will receive usual care as provided within their home.

INTERVENTIONS:
Behavioral: PREVENT Program — A standardized PREVENT educational program will be offered to each intervention LTC home and health-care staff. The curricula includes video modules with fracture-prevention care recommendations and an orientation to the Fracture Prevention Toolkit. Using the Fracture Risk Scale (i.e., a clinical decision support tool embedded in the RAI-MDS 2.0), the LTC team will identify residents at high-risk for fracture and will implement the fracture prevention recommendations into care plans on an individual resident basis.
  Arms: PREVENT Program

SUMMARY:
Hip fractures occur nearly twice as often for older adults residing in long-term care as they do in older adults of a similar age still living in other settings. Hip fractures are the leading cause of hospitalization and often result in loss of independence, problems with walking and sometimes death. To address this problem the PREVENT (Person-centered Routine Fracture PrEVENTion in LTC) program was designed for use in long-term care homes. PREVENT uses a tool ("fracture risk calculator") based on a residents electronic health record to capture who is most at risk of fracture due to osteoporosis and falls. The program then trains the health care team including doctors, pharmacists and nurses on the latest recommendations on how to best assist residents and their families in making treatment decisions. The healthcare teams are also given tools that help them stay on track such as templates for ordering medications, strategies to reduce falls and fractures and making care plans. The study will examine if this program is effective for decreasing hip fractures by assigning some homes to receive the PREVENT program (intervention group) and some homes to usual care (control group) and comparing the results.

ELIGIBILITY:
Inclusion Criteria:

* Both profit and non-profit long-term care homes in Ontario, Canada.
* Homes must have a minimum of 50 occupied beds to participate; there is no maximum home size for participation.
* For both control and intervention homes, resident eligibility (and study cohorts) will be determined via the RAI-MDS 2.0 database.

Exclusion Criteria:

* Residents identified as having end-stage disease, who are comatose, receiving hospice or respite care and who have an expected short stay (90 days or less).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3060 (Estimated)
Dates: Start 2024-06-19 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of hip-fractures | One year
  Data extracted from the Discharge Abstract Database (DAD) and National Ambulatory Care Reporting System (NACRS). Scored as occurred: yes, no.

SECONDARY OUTCOMES:
Number of non-hip fractures (wrist, spine, pelvis, humerus) | One year
  Data extracted from the DAD and NACRS datasets. Scored as occurred: yes, no.
Number of hospital transfers (emergency department and admissions) | One year
  Data extracted from the DAD and NACRS datasets. Scored as occurred: yes, no.
Number of deaths | One year
  Data extracted from the DAD and NACRS datasets. Scored as occurred: yes, no.
Change in number of falls | Baseline, 3, 6, 9 and 12 months
  Assessed by the Minimum Data Set (MDS) (standardized assessment) 2.0. Scored as occurred: yes, no and number of falls.
Change in level of pain | Baseline, 3, 6, 9 and 12 months
  Assessed by the MDS 2.0 Pain Scale. Scored on a scale from 0-4 where higher scores indicate more severe pain.
Change in mobility | Baseline, 3, 6, 9 and 12 months
  Assessed by the MDS 2.0 Activities of Daily Living (ADL) Hierarchy Scale. Scored on a scale from 0-6 where higher scores indicate more impairment in ADL performance.
Change in responsive behaviours | Baseline, 3, 6, 9 and 12 months
  Assessed by the MDS 2.0 Aggressive Behaviour Scale. Scored on a scale from 0-12 where higher scores indicate greater frequency and diversity of aggressive behaviour.
Change in health related quality of life | Baseline, 3, 6, 9 and 12 months
  Assessed by the MDS 2.0 Health Status Index. Scored on a scale from 0-1 where a score of 1 indicates full health.
Change in medications | Baseline, 3, 6, 9 and 12 months
  Data extracted from the pharmacy database. Recorded as number of LTC residents receiving osteoporosis medication(s).
Health quality indicators | Baseline, 3, 6, 9 and 12 months.
  Assessed by the Minimum Data Set (MDS) (standardized assessment) 2.0 or health quality indicators for falls, pressure ulcers, pain, physical function and depression.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Papaioannou, MD, MSc, Principal Investigator — McMaster University
Locations (1):
- McMaster University - St. Peter's Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Papaioannou A, Feldman S, Katz P, Costa AP, Kennedy CC, Adachi JD, Boyd H, Giangregorio L, Heckman G, Hewston P, Hirdes J, Holroyd-Leduc J, Howard M, Ho J, Jaglal S, Kaasalainen S, Kristof L, Lau A, Lee J, McArthur C, Marr S, O'Donnell D, Rodrigues IB, Shankardass K, Siu H, Straus S, Thrall S, Tarride JE, Thabane L, Hafid S, Tung J, Hillier LM, Kane LL, Azizudin AM, Desinghe TD, Ioannidis G. Study protocol for a pragmatic, cluster, randomized controlled trial of a multifaceted fracture prevention model for long-term care: the PREVENT trial. Trials. 2026 Jan 9;27(1):111. doi: 10.1186/s13063-025-09398-1. PMID 41507969